CLINICAL TRIAL: NCT00049439
Title: Dose-Modified Oral Combination Chemotherapy In Patients With Aids-Related Non-Hodgkin's Lymphoma In The United States And Africa
Brief Title: Combination Chemotherapy in Treating Patients With AIDS-Related Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensvie Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2498; P30CA043703 (NIH); CWRU-029828J; CWRU-2498; NCI-G02-2126; CASE-2498
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma
Keywords: AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related small noncleaved cell lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Filgrastim; Cyclophosphamide; Etoposide; Lomustine; Procarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — filgrastim (G-CSF) subcutaneously on days 5-21 and 28-42. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
Drug: cyclophosphamide — Oral cyclophosphamide on days 22-26. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
Drug: etoposide — Oral etoposide on days 1-3. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
Drug: lomustine — Oral lomustine on day 1 (course 1 only). Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
Drug: procarbazine hydrochloride — Oral procarbazine on days 22-26. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining lomustine, etoposide, cyclophosphamide, and procarbazine in treating patients who have AIDS-related non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate, response duration, and survival of patients with AIDS-related non-Hodgkin's lymphoma treated with lomustine, etoposide, cyclophosphamide, and procarbazine.
* Determine the feasibility of this regimen in these patients.
* Determine the clinical toxicity of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.
* Determine the impact of this regimen on the underlying HIV infection in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral lomustine on day 1 (course 1 only), oral etoposide on days 1-3, and oral cyclophosphamide and oral procarbazine on days 22-26. Patients may also receive filgrastim (G-CSF) subcutaneously on days 5-21 and 28-42. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on days 1 and 22 of each course, at day 84, and then every 3 months for 1 year.

Patients are followed at day 84 and then every 3 months.

PROJECTED ACCRUAL: A total of 66 patients (22 in the United States and 44 in Africa) will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acquired immune deficiency syndrome
* Histologically confirmed stage I, II, III, or IV intermediate- or high-grade non-Hodgkin's lymphoma

  * B-cell, T-cell, or indeterminate immunologic phenotype
* Measurable or evaluable disease
* No clinical, radiographic, or cytological evidence of CNS parenchymal, vitreal, or leptomeningeal involvement by lymphoma NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over (in the United States)
* 16 and over (in Africa)

Performance status

* ECOG 0-3

Life expectancy

* At least 6 weeks

Hematopoietic

* WBC at least 1,500/mm3
* Platelet count at least 50,000/mm3

Hepatic

* Bilirubin no greater than 3.0 mg/dL

Renal

* Creatinine no greater than 3.0 mg/dL

Other

* Concurrent active infection for which patient is receiving treatment allowed provided clinical status is stable
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for lymphoma

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy for stage I or II disease allowed provided there is documentation of disease progression

Surgery

* Not specified

Other

* Concurrent antiretroviral therapy (except zidovudine) allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1998-03; Primary Completion 2005-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Disease response | Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

SECONDARY OUTCOMES:
Quality of life as assessed by the Functional Living Index-Cancer and the Brief Symptom Inventory | days 1 and 2 of courses 1 and 2 and on day 84

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (4):
- United States (2):
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
- University of Nairobi College of Health Sciences, Nairobi, Kenya
- Uganda Cancer Institute, Kampala, Uganda